CLINICAL TRIAL: NCT02844530
Title: Randomized Phase II Study Evaluating the Efficacy of 90Yttrium-epratuzumab Tetraxetan Radioimmunotherapy in Adults With CD22+ Relapsed/Refractory B-ALL
Brief Title: Study Evaluating the Efficacy of 90Yttrium-epratuzumab in Adults With CD22+ Relapsed/Refractory B-ALL
Acronym: RITEPRALL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC15_0088
Record Dates: First submitted 2015-11-13; First posted 2016-07-26 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: CD22+ Relapsed/Refractory B-ALL
Keywords: adults
MeSH Terms: interventions — Drug Therapy; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIT (Experimental): The experimental treatment will consist on 2 injections of 370 MBq/m2 of 90Y-epratuzumab tetraxetan fractionated RIT at day 1 and day 8. The first infusion of 90Y-epratuzumab tetraxetan will be co-injected for the six first patients in Nantes with 111In-epratuzumab tetraxetan for dosimetry purpose.
  Interventions: Drug: 90Y-epratuzumab tetraxetan
- chemotherapy/ immunotherapy (Active Comparator): chemotherapy/ immunotherapy regimen will be assigned per investigator's choice to one of the following chemotherapy/ immunotherapy regimens:
  1. FLAG +- anthracycline based regimen For subject's >60 years : idarubicin 5 mg/m2 day 1,3, fludarabine 20 mg/m2 days 1-5, cytarabine 1 g/m2 days 1-5.
  2. Clofarabine or clofarabine based regimens. Clofarabine use as a single agent should follow the recommended prescribing information. Clofarabine combination based regimens should use >=20mg/m2/day for up to 5 days.
  3. Hyper-C-VAd regimen: hyperfractionated cyclophosphamide 300 mg/m2 intravenously(i.v.) every 12 hours for 6 doses Days 1 to 3 + vincristine 2 mg i.v.Days 4 and 11; doxorubicin 50 mg/m2 i.v. over 24 hours via central venous catheter Day 4; and dexa-methasone 40 mg daily Days 1 to 4 and 11 to 14.
  4. Blinatumomab (Blincyto®) : 28-day continuous infusion (9µg/d for days 1-7; 28µg/d thereafter, followed by 2 weeks of rest for up to 2 cycles.
  Interventions: Drug: chemotherapy/ immunotherapy

INTERVENTIONS:
Drug: 90Y-epratuzumab tetraxetan — The Primary objective is to compare the complete response rate (CR + CRp) after 2 injections of 370 MBq/m² of 90Y-epratuzumab tetraxetan RIT at day 1 and day 8 versus standard of care salvage chemotherapy regimens in adult CD22+ relapsed/refractory B-ALL.
  A second RIT cycle (consolidation) will be allowed in the experimental group in case of response (CR or CRp).
  From an ethical point of view, it will be also permitted to propose the RIT experimental treatment in the control group in case of treatment failure or relapse during the 6 months following inclusion. Follow-up will be also 12 months from the RIT for these patients
  Other Names: 90Y-DOTA-hLL2 or 90Y-DOTA-Epratuzumab
  Arms: RIT
Drug: chemotherapy/ immunotherapy
  Arms: chemotherapy/ immunotherapy

SUMMARY:
The investigators propose a randomized phase 2 study evaluating 90Y-epratuzumab tetraxetan for relapsed/refractory CD22+ B-ALL adult patients using the recommended activity of 370 MBq/m² x 2. in order to confirm the investigators' previous results. The cut-off of 70% for the expression of CD22 has been chosen in order to propose this protocol to all adults with CD22+ B ALL in relapse or with refractory disease. Indeed, median expression of CD22 is almost 100% in this setting but some patients are documented between 70 and 100%. RIT will be assessed in comparison with standard of care salvage chemotherapy regimens. Only three standard salvage chemotherapy regimens will be permitted in order to avoid too much bias for the comparative analysis of clinical efficacy.

DETAILED DESCRIPTION:
The experimental treatment will consist on 2 injections of 370 MBq/m2 of 90Y-epratuzumab tetraxetan fractionated RIT at day 1 and day 8. The first infusion of 90Y-epratuzumab tetraxetan will be co-injected for the six first patients in Nantes with 111In-epratuzumab tetraxetan for dosimetry purpose.

Subjects randomized to receive standard of care salvage chemotherapy/ immunotherapy regimen will be assigned per investigator's choice to one of the following chemotherapy/ immunotherapy regimens:

1. FLAG +- anthracycline based regimen (such as Idarubicin 10 mg/m2 days 1, 3; fludarabine 30 mg/m2 days 1-5, cytarabine 2 g/m2 days 1-5).

   For subject's >60 years : idarubicin 5 mg/m2 day 1,3, fludarabine 20 mg/m2 days 1-5, cytarabine 1 g/m2 days 1-5.
2. Clofarabine or clofarabine based regimens. Clofarabine use as a single agent should follow the recommended prescribing information. Clofarabine combination based regimens should use >=20mg/m2/day for up to 5 days.
3. Hyper-C-VAd regimen: hyperfractionated cyclophosphamide 300 mg/m2 intravenously(i.v.) every 12 hours for 6 doses Days 1 to 3 + vincristine 2 mg i.v.Days 4 and 11; doxorubicin 50 mg/m2 i.v. over 24 hours via central venous catheter Day 4; and dexa-methasone 40 mg daily Days 1 to 4 and 11 to 14.
4. Blinatumomab (Blincyto®) is administered as a 28-day continuous infusion (9µg/d for days 1-7; 28µg/d thereafter, followed by 2 weeks of rest for up to 2 cycles. Patients should be hospitalized the first 9 days during the first cycle and at least the first 2 days during the second cycle.

A second RIT cycle (consolidation) will be allowed in the experimental group in case of response (CR or CRp).

From an ethical point of view, it will be also permitted to propose the RIT experimental treatment in the control group in case of treatment failure or relapse during the 6 months following inclusion. Follow-up will be also 12 months from the RIT for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age>= 18 years old
* Philadelphia positive or negative B-ALL (OMS) with >5% of blasts in bone marrow with or without extramedullary disease
* CD22+ expression >=30% of the blast population
* Refractory B-ALL defined by :

  * treatment failure after 1 or 2 successive courses of induction therapy or first relapse <6 months from CR.
  * First relapse, second or third relapse.
  * Unresponsive to prior treatment with >=1 second/third (dasatinib, nilotinib, bosutinib, ponatinib) generation TKIs and standard induction chemotherapy for Ph+ B-ALL patients only.
* Peripheral absolute lymphoblast count <10000/µL: hydroxyurea and/or steroids/vincristine treatment within 2 weeks of randomization is allowed to reduce circulating blasts.
* ECOG (Eastern Cooperative Oncology Group) < 2
* Creatinine clearance >= 50 ml/min (Cockroft formula) or serum creatinine <=1.5 x ULN
* Adequate hepatic function: total serum bilirubin < 1.5 x upper limit of normal (ULN) except for documented Gilbert syndrome or considered tumor related; <=5 ULN for transaminases except if considered tumor related
* Written informed consent
* Having or not received previously Epratuzumab: in case of having received previously epratuzumab, patients should be free of HAHA (anti-epratuzumab antibodies).
* Patient affiliated to or beneficiary of the National Health Service
* Patients with lymphoblastic lymphoma can be included if they satisfied all eligibility criteria.

Non-inclusion criteria:

* T-ALL, patients with Burkitt lymphoma
* Active Meningeal involvement
* Isolated extramedullary relapse
* CD22 expression on tumor cells or < 30%
* HIV positive
* Active Hepatitis B or C
* Allogeneic transplantation within 12 weeks prior to the start of chemo/immunotherapy or RIT
* Active acute or chronic GVHD, systemic treatment of GVHD within two weeks before the treatment start.
* No chemotherapy/immunotherapy <2 weeks before randomization except to reduce the circulating lymphoblast count.
* Left ventricular ejection fraction < 45%
* Contra-indication to 90Y-epratuzumab tetraxetan
* Previous or concurrent second malignancy except for adequately treated basal cell carcinoma of the skin, curatively treated in situ carcinoma of the cervix, curatively treated solid cancer, with no evidence of disease for at least 2 years
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Participation at the same time in another study in which investigational drugs are used
* Absence of written informed consent
* Pregnant or breastfeeding women
* Women or men without effective contraceptive barrier if needed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Compare the complete response rate (CR + CRp) in the two arms | Week 4 to Week 6
  Evaluated between 4 and 6 weeks from day 1. Blood and bone marrow analysis.

SECONDARY OUTCOMES:
Overall survival: overall and comparison between both groups | Month 1 to Month 12
  clinical follow up
Disease free survival | Month 1 to Month 12
  clinical follow up
time to disease progression | Month 1 to Month 12
  clinical follow up
duration of response | Month 1 to Month 12
  clinical follow up
CD22 expression | Month 1 to Month 12
  bone marrow analysis
CD22 expression | Month 1 to Month 12
  blood
Safety and tolerance of fractionated RIT with 90Y-epratuzumab tetraxetan assessed by NCI Criteria | Month 1 to Month 12
  NCI Criteria
Immunization test to search for antibodies by ELISA test | Month 1 to Month 6
  Blood assay (ELISA method)
Realization of a blood pharmacokinetics profile of 111In /90Y-epratuzumab tetraxetan | 1 week after 90Y-epratuzumab tetraxetan injection
  Blood counting
Tumour and organ dosimetry of 90Y-epratuzumab tetraxetan assessed using 111In-epratuzumab tetraxetan biodistribution | 1 week after 90Y-epratuzumab tetraxetan injection
  dosimetry analysis
Correlation between FLT3-ligand serum value and efficacy and toxicity after treatment | Month 1 to Month 12
  Blood analysis
Relapse incidence: overall and comparison between both groups | Month 1 to Month 12
  blood
Relapse incidence: overall and comparison between both groups | Month 1 to Month 12
  bone marrow analysis
Minimal Residual Disease (MRD) (by FACS analysis) | Month 1 to Month 12
  blood
Minimal Residual Disease (MRD) (by FACS analysis) | Month 1 to Month 12
  bone marrow analysis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France